CLINICAL TRIAL: NCT06600750
Title: Artificial Intelligence-based Prediction of Radio-cephalic Arteriovenous Fistula Maturation Using Preoperative Duplex Examination
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ara Cho, Professor, Seoul National University Hospital
Other Study IDs: S2020-3118-0001
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Renal Insufficiency, Chronic; Arteriovenous Fistula; Artificial Intelligence (AI); Machine Learning
Keywords: Preoperative Ultrasound Mapping; Radiocephalic Arteriovenous Fistula; Renal Dialysis; Artificial intelligence; Machine Learning; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula | interventions — Arteriovenous Shunt, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who underwent radiocephalic arteriovenous fistula due to advanced chronic kidney disease: Patients who underwent radiocephalic arteriovenous fistula due to advanced chronic kidney disease
  Interventions: Procedure: Arteriovenous fistula

INTERVENTIONS:
Procedure: Arteriovenous fistula — Patients who underwent Radiocephalic arteriovenous fistula surgery

SUMMARY:
The goal of this observational study is to assess the efficacy of AI-driven models in analyzing comprehensive ultrasonographic variables across multiple forearm locations to predict successful AVF maturation. The main question it aims to answer is:

Can AI-driven models analyzing comprehensive ultrasonographic variables accurately predict the successful maturation of arteriovenous fistulas (AVFs)?

Participants who underwent radiocephalic arteriovenous fistula (AVF) creation had their preoperative ultrasonographic data analyzed using AI-driven models to predict successful AVF maturation over a four-year retrospective period.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent RCAVF due to advanced chronic kidney disease from 2018 to 2022

Exclusion Criteria:

* Patients who did not have follow-up data available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent RCAVF due to advanced chronic kidney disease from 2018 to 2022
Sampling Method: Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Maturation of the fistula | 90 days
  Fistula maturation was defined as an arteriovenous fistula that matures and is usable for dialysis with two-needle cannulation for hemodialysis for at least 90 days without the need for endovascular or surgical interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Georgiadis GS, Charalampidis DG, Argyriou C, Georgakarakos EI, Lazarides MK. The Necessity for Routine Pre-operative Ultrasound Mapping Before Arteriovenous Fistula Creation: A Meta-analysis. Eur J Vasc Endovasc Surg. 2015 May;49(5):600-5. doi: 10.1016/j.ejvs.2015.01.012. Epub 2015 Feb 27. PMID 25736517
- [Background] Vascular Access Work Group. Clinical practice guidelines for vascular access. Am J Kidney Dis. 2006 Jul;48 Suppl 1:S248-73. doi: 10.1053/j.ajkd.2006.04.040. No abstract available. PMID 16813991
- [Background] Perera GB, Mueller MP, Kubaska SM, Wilson SE, Lawrence PF, Fujitani RM. Superiority of autogenous arteriovenous hemodialysis access: maintenance of function with fewer secondary interventions. Ann Vasc Surg. 2004 Jan;18(1):66-73. doi: 10.1007/s10016-003-0094-y. Epub 2004 Jan 20. PMID 14727162